CLINICAL TRIAL: NCT00557726
Title: Diagnosis and Management of Inflammatory and Infectious Diseases
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 780023; 78-I-0023
Record Dates: First submitted 2007-11-10; First posted 2007-11-14 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-04-16

CONDITIONS: Infection; Inflammation
Keywords: Inflammation; Infection; Fever; Natural History
MeSH Terms: conditions — Infections; Inflammation; Fever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients with a variety of infections and inflammatory diseases.

SUMMARY:
This protocol is being established to cover the evaluation of patients with inflammatory and/or infectious diseases which are not covered under previously existing protocols. The purpose of such a protocol is that frequently patients are referred to us with either diagnosed or undiagnosed illnesses which would be of interest to our teaching program or which would serve as a source of patients to subsequently be entered into established, ongoing protocol studies. Such patients will be admitted to the protocol and handled according to accepted medical practice of diagnosis and treatment.

DETAILED DESCRIPTION:
Study Description:

This protocol was established in 1978 to evaluate patients with diagnosed and undiagnosed inflammatory and/or infectious diseases that are of scientific interest. Once diagnosis is made patients are referred to relevant NIH protocols for follow-up. If an NIH protocol does not exist for the condition, participants receive the required clinical standard of care treatment through an outside provider or through this protocol if a provider with the necessary expertise cannot be found. It is a minimal risk study.

Objective:

To evaluate patients with possible infectious and/or inflammatory diseases in order to collect data/samples through the diagnosis of infectious and inflammatory conditions (including in terms of clinical, immunologic, and metabolic features) further characterize, and treat infectious and inflammatory conditions through the collection of clinical specimens, medical records and in-person assessments

To provide a repository of information on enrolled participants to allow for hypothesis generation in future research

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Known or suspected exposure to infection, as determined by the Principal Investigator OR Presence of signs and symptoms of an infectious or inflammatory disease
  2. Age range: 3 years of age and older.
  3. NIAID/LIR investigator who has an interest in the patient s illness and is willing to serve as attending physician to supervise the patient's medical care at the NIH.
  4. Primary physician outside the NIH
  5. The patient or the patient's Legally Authorized Representative is capable of informed consent and signs the consent form. The consent form will be signed by parents or guardians of patients under the age of 18

EXCLUSION CRITERIA:

1. Pregnant.
2. Presence of conditions that, in the judgment of the investigator, may put the participant at undue risk or make them unsuitable for participation in the study.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with an inflammatory or infectious condition are evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 1978-02-17 (Actual)

PRIMARY OUTCOMES:
H&P, labs and other clinical metrics | initial and follow-up clinic visits
  this is a hypothesis-generating training consult protocol

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Wright, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual results and Physician's notes will be shared with Primary Care Providers as identified by the study participant.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1978-I-0023.html